CLINICAL TRIAL: NCT07216664
Title: Randomized Controlled Trial of Multisensory Early Oral Administration of Human Milk (M-MILK) for Very Preterm Infants: Enhancing Stress Regulation, Neurodevelopment, and Oral Feeding Skills
Brief Title: Multisensory Early Oral Administration of Human Milk (M-MILK) for Very Preterm Infants
Acronym: M-MILK RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 218601
Record Dates: First submitted 2024-09-26; First posted 2025-10-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-MILK Group (Experimental): Infants in the M-MILK group will receive M-MILK intervention and standard of care. M-MILK is implemented starting on day 3 of life, during the day shift, after every hands-on care, during the beginning of a full gavage feeding, and up to 4 times a day. Infants receive M-MILK in small droplets via a 1-ml syringe. M-MILK will cease upon oral feeding initiation. Infants will receive either mother's own milk or donor's milk based on availability. Infants may receive up to 1 mL of milk each time based on their cues and responses. The 1 mL volume intake is included as part of their oral caloric intake. M-MILK is provided by research nurses or parents.
  Interventions: Other: Multisensory early oral administration of human milk
- Control Group (No Intervention): Infants in the Control group will receive standard of care.

INTERVENTIONS:
Other: Multisensory early oral administration of human milk — M-MILK is implemented starting on day 3 of life, during the day shift, after every hands-on care, during the beginning of a full gavage feeding, and up to 4 times a day. Infants receive M-MILK in small droplets via a 1-ml syringe. M-MILK will cease upon oral feeding initiation. Infants will receive either mother's own milk or donor's milk based on availability. Infants may receive up to 1 mL of milk each time based on their cues and responses. The 1 mL volume intake is included as part of their oral caloric intake. M-MILK is provided by research nurses or parents.
  Other Names: M-MILK
  Arms: M-MILK Group

SUMMARY:
The goal of this clinical trial is to learn if the multisensory early oral administration of human milk (M-MILK) intervention helps infants who are born younger than 32 weeks gestational age (very preterm infants). The main question that this clinical trial aims to answer is: Does M-MILK improve stress regulation, support optimal neurodevelopment, and promote competent oral feeding skills in very preterm infants?

Researchers will compare M-MILK to the standard of care to see if M-MILK helps very preterm infants. Specifically, researchers will compare the differences in:

* Cortisol levels
* DNA methylation of the two stress related genes (NR3C1 and HSD11B2)
* Neurodevelopment
* Oral feeding skills Participants in the M-MILK group will receive standard of care plus M-MILK intervention, which starts on day 3 of life and continues until they begin their oral feeding. M-MILK will be provided by clinical research nurses, during the day shift, up to 4 times a day. Participants in the standard of care group will continue to receive their usual care.

ELIGIBILITY:
Inclusion Criteria:

* Born at ≤ 32 weeks gestational age.
* Receiving mother's own milk and/or donor human milk at the time of screening.

Exclusion Criteria:

* Receiving only formula.
* Gastrointestinal defects, i.e., cleft lip or cleft palate.
* Congenital cardiac defects requiring surgery.
* Necrotizing enterocolitis.
* Chromosomal abnormalities.

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Oral feeding Skills: EFS assessment total score at PO Initiation | Up to 12 weeks after birth.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at oral feeding (PO) initiation. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment total score at 36 Weeks PMA | 36 weeks postmenstrual age.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at 36 weeks post-menstrual age (PMA). The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.

SECONDARY OUTCOMES:
Stress Regulation: Salivary Cortisol at PO Initiation | Up to 12 weeks after birth.
  We will evaluate stress regulation, measured by salivary cortisol levels (μg/dL) at oral feeding (PO) initiation.
Stress Regulation: Salivary Cortisol at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate stress regulation, measured by salivary cortisol levels (μg/dL) at 36 weeks PMA.
Stress Regulation: Buccal Cell DNAm of NR3C1 Exon 1F Promoter at PO Initiation | Up to 12 weeks after birth.
  We will evaluate stress regulation, measured by buccal cell DNA methylation (DNAm) of NR3C1 Exon 1F promoter at oral feeding (PO) initiation. We anticipate to cover 33 CpG sites within the NR3C1 Exon 1F promoter. Methylation percentage (%) will calculated per CpG site (aligning with the human reference genome hg38).
Stress Regulation: Buccal Cell DNAm of NR3C1 Exon 1F Promoter at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate stress regulation, measured by buccal cell DNA methylation (DNAm) of NR3C1 Exon 1F promoter at 36 weeks post-menstrual age (PMA). We anticipate to cover 33 CpG sites within the NR3C1 Exon 1F promoter. Methylation percentage (%) will calculated per CpG site (aligning with the human reference genome hg38).
Stress Regulation: Buccal Cell DNAm of HSD11B2 Promoter at PO Initiation | Up to 12 weeks after birth.
  We will evaluate stress regulation, measured by buccal cell DNA methylation (DNAm) of HSD11B2 promoter at oral feeding (PO) initiation. We anticipate to cover 30 CpG sites within the HSD11B2 promoter. Methylation percentage (%) will calculated per CpG site (aligning with the human reference genome hg38).
Stress Regulation: Buccal Cell DNAm of HSD11B2 Promoter at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate stress regulation, measured by buccal cell DNA methylation (DNAm) of HSD11B2 promoter at 36 weeks post-menstrual age (PMA). We anticipate to cover 30 CpG sites within the HSD11B2 promoter. Methylation percentage (%) will calculated per CpG site (aligning with the human reference genome hg38).
Neurodevelopment: NNNS-II Attention score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Handling score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Self-Regulation 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Habituation score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Arousal score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Excitability score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Lethargy score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Hypertonicity score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Hypotonicity score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Nonoptimal Reflexes score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Asymmetric Reflexes score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Quality of Movement score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.
Neurodevelopment: NNNS-II Stress/Abstinence score 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate neurodevelopment using the NeoNatal Neurobehavioral Scale (NNNS-II) at 36 weeks post-menstrual age (PMA). The NNNS-II provides a summary score for each of the 13 domain (attention, handling, self-regulation, habituation, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, quality of movement, and stress/abstinence). High-risk neurodevelopment is characterized by higher scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence, along with lower score in quality of movement, attention, self-regulation, habituation. Low-risk neurodevelopment is characterized by higher scores in attention, self-regulation, habituation, and quality of movement, along with lower scores in handling, arousal, excitability, lethargy, hypertonicity, hypotonicity, nonoptimal reflexes, asymmetric reflexes, and stress/abstinence.

OTHER OUTCOMES:
Oral Feeding Skills: EFS assessment score for Respiratory Regulation at PO Initiation | Up to 12 weeks after birth.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at oral feeding (PO) initiation. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Oral-motor Functioning at PO Initiation | Up to 12 weeks after birth.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at oral feeding (PO) initiation. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Swallowing Coordination at PO Initiation | Up to 12 weeks after birth.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at oral feeding (PO) initiation. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Engagement at PO Initiation | Up to 12 weeks after birth.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at oral feeding (PO) initiation. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Physiologic Stability at PO Initiation | Up to 12 weeks after birth.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at oral feeding (PO) initiation. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Respiratory Regulation at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at 36 weeks PMA. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Oral-motor Functioning at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at 36 weeks PMA. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Swallowing Coordination at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at 36 weeks PMA. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Engagement at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at 36 weeks PMA. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: EFS assessment score for Physiologic Stability at 36 Weeks PMA | At 36 weeks postmenstrual age.
  We will evaluate oral feeding skills using the Early Feeding Skills Assessment (EFS) at 36 weeks PMA. The EFS provides a summary score for each of the 5 subscale (respiratory regulation, oral-motor functioning, swallowing coordination, engagement, and physiologic stability), as well as a total summary score. Higher EFS summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: NeoEAT Total score at 2 Months CA | At 2 months corrected age.
  We will evaluate oral feeding skills using the Neonatal Eating Assessment Tool (NeoEAT-Bottle-feeding) at 2 months corrected age (CA). The NeoEAT-Bottle-feeding provides a summary score for each of the 5 subscale (regulation, energy and physiologic stability, gastrointestinal tract function, sensory responsiveness, and compelling symptoms of problematic feeding) and a total summary score. Lower NeoEAT-Bottle-feeding summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: NeoEAT score for Regulation at 2 Months CA | At 2 months corrected age.
  We will evaluate oral feeding skills using the Neonatal Eating Assessment Tool (NeoEAT-Bottle-feeding) at 2 months corrected age (CA). The NeoEAT-Bottle-feeding provides a summary score for each of the 5 subscale (regulation, energy and physiologic stability, gastrointestinal tract function, sensory responsiveness, and compelling symptoms of problematic feeding) and a total summary score. Lower NeoEAT-Bottle-feeding summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: NeoEAT score for Energy and Physiologic Stability at 2 Months CA | At 2 months corrected age.
  We will evaluate oral feeding skills using the Neonatal Eating Assessment Tool (NeoEAT-Bottle-feeding) at 2 months corrected age (CA). The NeoEAT-Bottle-feeding provides a summary score for each of the 5 subscale (regulation, energy and physiologic stability, gastrointestinal tract function, sensory responsiveness, and compelling symptoms of problematic feeding) and a total summary score. Lower NeoEAT-Bottle-feeding summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: NeoEAT score for Gastrointestinal Tract Function at 2 Months CA | At 2 months corrected age.
  We will evaluate oral feeding skills using the Neonatal Eating Assessment Tool (NeoEAT-Bottle-feeding) at 2 months corrected age (CA). The NeoEAT-Bottle-feeding provides a summary score for each of the 5 subscale (regulation, energy and physiologic stability, gastrointestinal tract function, sensory responsiveness, and compelling symptoms of problematic feeding) and a total summary score. Lower NeoEAT-Bottle-feeding summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: NeoEAT score for Sensory Responsiveness at 2 Months CA | At 2 months corrected age.
  We will evaluate oral feeding skills using the Neonatal Eating Assessment Tool (NeoEAT-Bottle-feeding) at 2 months corrected age (CA). The NeoEAT-Bottle-feeding provides a summary score for each of the 5 subscale (regulation, energy and physiologic stability, gastrointestinal tract function, sensory responsiveness, and compelling symptoms of problematic feeding) and a total summary score. Lower NeoEAT-Bottle-feeding summary scores indicate more competent oral feeding skills.
Oral Feeding Skills: NeoEAT score for Compelling Symptoms of Problematic Feeding at 2 Months CA | At 2 months corrected age.
  We will evaluate oral feeding skills using the Neonatal Eating Assessment Tool (NeoEAT-Bottle-feeding) at 2 months corrected age (CA). The NeoEAT-Bottle-feeding provides a summary score for each of the 5 subscale (regulation, energy and physiologic stability, gastrointestinal tract function, sensory responsiveness, and compelling symptoms of problematic feeding) and a total summary score. Lower NeoEAT-Bottle-feeding summary scores indicate more competent oral feeding skills.
Neurodevelopment: ASQ-3 Communication score at 2 Months CA | At 2 months corrected age.
  We will evaluate neurodevelopment using the Ages and Stages Questionnaire (ASQ-3) at 2 months corrected age (CA). The 2-month ASQ-3 provides a summary score for each of the 3 domain (communication, gross motor, and personal-social skills). Higher summary scores indicate more optimal neurodevelopment.
Neurodevelopment: ASQ-3 Gross Motor score at 2 Months CA | At 2 months corrected age.
  We will evaluate neurodevelopment using the Ages and Stages Questionnaire (ASQ-3) at 2 months corrected age (CA). The 2-month ASQ-3 provides a summary score for each of the 3 domain (communication, gross motor, and personal-social skills). Higher summary scores indicate more optimal neurodevelopment.
Neurodevelopment: ASQ-3 Personal-Social Skills score at 2 Months CA | At 2 months corrected age.
  We will evaluate neurodevelopment using the Ages and Stages Questionnaire (ASQ-3) at 2 months corrected age (CA). The 2-month ASQ-3 provides a summary score for each of the 3 domain (communication, gross motor, and personal-social skills). Higher summary scores indicate more optimal neurodevelopment.

CONTACTS AND LOCATIONS:
Overall Officials: Thao Griffith, PhD, Principal Investigator — Loyola University Chicago
Locations (2):
- United States (2):
  - Loyola University Chicago, Maywood, Illinois
  - Loyola University Medical Center, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD to ensure confidentiality and privacy participants. We have plans to share only de-identifiable data. Data will be shared in accordance with the NIH Data Sharing Policy. Data will be shared on reasonable request to Loyola University Chicago through a Data Use Agreement (DUA).

REFERENCES:
- [Derived] Griffith T, Janusek L, White-Traut R, Green SJ, Sachin A, Joyce C. Study Protocol for a Randomized Controlled Trial of Multisensory Early Oral Administration of Human Milk (M-MILK) for Very Preterm Infants: Enhancing Stress Regulation, Neurodevelopment, and Oral Feeding Skills. Biol Res Nurs. 2026 Jan 19:10998004261418708. doi: 10.1177/10998004261418708. Online ahead of print. PMID 41554032